CLINICAL TRIAL: NCT01750775
Title: Shensongyangxin Capsule in the Treatment of Sinus Bradycardia With Premature Ventricular Contractions Multi-center,Randomized, Double-blind, Placebo-controlled Clinical Study
Brief Title: Shensongyangxin Capsule in the Treatment of Sinus Bradycardia With Premature Ventricular Contractions
Acronym: SS-SBVPT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: kejiang Cao (Other)
Collaborators: Chinese Academy of Medical Sciences, Fuwai Hospital (Other); Third Military Medical University (Other)
Responsible Party: Sponsor-Investigator, kejiang Cao, director of cardiology cepartment, The First Affiliated Hospital with Nanjing Medical University
Organization: The First Affiliated Hospital with Nanjing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: yl-yxb07-lcsyfa-201202; ChiCTR-TRC-12002504 (Other: ChiCTR)
Record Dates: First submitted 2012-12-06; First posted 2012-12-17 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Premature Ventricular Contraction
Keywords: sinus bradycardia; ventricular premature contraction
MeSH Terms: conditions — Ventricular Premature Complexes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Shensong Yangxin capsule (Experimental): Shensong Yangxin capsule 4 granules t.i.d. by mouth for 8weeks
  Interventions: Drug: Shensong Yangxin capsule
- placebo Capsule (Placebo Comparator): placebo Capsule 4 granules t.i.d. by mouth for 8 weeks
  Interventions: Drug: placebo Capsule

INTERVENTIONS:
Drug: Shensong Yangxin capsule — ShenSongYangXin Capsule 4 granules t.i.d. by mouth for 8 weeks
  Arms: Shensong Yangxin capsule
Drug: placebo Capsule — placebo Capsule 4 granules t.i.d. by mouth for 8 weeks
  Arms: placebo Capsule

SUMMARY:
The purpose of this study is to assess the effects of Chinese medicine Shansong Yangxin capsule for sinus bradycardia complicated with ventricular premature beats.

DETAILED DESCRIPTION:
Premature ventricular contractions is one of the most common symptomatic arrhythmia. Antiarrhythmia drugs for premature ventricular contractions, such as beta-blockers and sodium channel blockers, can cause bradycardia. For sinus bradycardia patients complicated with premature ventricular contractions, it's hard for doctors to make decision. The purpose of the study is to assess the effects of Chinese medicine Shansong Yangxin capsule for sinus bradycardia complicated with ventricular premature beats, which based on the numbers of premature ventricular contractions and average hear rate in 24-hour ambulatory electrocardiogram (ECG) after 8 weeks treatment as the primary endpoint of the study. Secondary endpoints are evaluation of the Shensong Yangxin capsule on quality of life. This study is a randomized, double-blind, placebo controlled, multi-center trial. Sinus bradycardia patients(average heart rate 45-59 beat per minute) associated with premature ventricular contractions (PVC number >10000 / 24h), are involved in the study. Patients are randomly assigned into Shensong Yangxin capsule group or placebo group, with the capsule administration of 4 granules t.i.d.for 8 weeks. 24-hour ambulatory ECG, are observed at baseline,4 weeks and 8 weeks after the intervention. The primary outcomes are the numbers of premature ventricular contractions and average heat rate in 24-hour ambulatory ECG, and the secondary outcomes is Minnesota living with heart failure questionnaire (MLHFQ).

ELIGIBILITY:
Inclusion Criteria:

* 18 Years to 70 Years old
* Documented sinus bradycardia with average heart rate at 45-59 by 24hours ambulatory EKG
* Ventricular premature beats: >1000 beats/24 hours

Exclusion Criteria:

* Younger than 18 years or older than 75 years
* Symptomatic sinus arrest >3 seconds or high degree atrioventricular block indicated for pacemaker
* Subject suffered from acute coronary syndrome in last three months (Acute myocardial infarction of ST segment elevation and non ST segment elevation, unstable angina
* To be complicated with persistent atrial fibrillation, or paroxysmal atrial fibrillation >5% during 24hrs ambulatory EKG or acute myocarditis
* To be complicated with ventricular fibrillation, torsion type ventricular heartbeat rate, sustained ventricular tachycardia, or non sustained ventricular tachycardia with rapid ventricular rate and hemodynamic disorders
* Sinus heart rate less than 45 beats/minutes and needs to receive the pacemaker or has received pacemaker, or with ICD,CRTP/D

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-09 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
numbers of the Premature ventricular contractions detected by 24 houres ambulatory EKG | 8 weeks
average heart rate detected by 24-hour ambulatory ECG | 8 weeks

SECONDARY OUTCOMES:
numbers of the Premature ventricular contractions detected by 24-hour ambulatory ECG | 4 weeks
average heart rate detected by 24-hour ambulatory ECG | 4 weeks

OTHER OUTCOMES:
Minnesota living with heart failure questionnaire (MLHFQ) | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kejiang Cao, M.D, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- the First Affiliated Hospital of Nanjing Medical Universtiy, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Zhang F, Zou J, Yu H, Li X, Kojodjojo P, Cai X, Zhang S, Huang C, Hong K, Yu B, Li G, Luo S, Zhou S, Zheng Y, Fan J, Cao X, Tao G, Sheng G, Bai Z, Jiang S, Liu X, Gu W, Chen F, Cao K. Acute Efficacy of a Traditional Chinese Medicine for Treatment of Frequent Premature Ventricular Contractions in Patients with Concomitant Sinus Bradycardia: Results from a Double-Blind, Placebo-Controlled, Multicentre, Randomized Clinical Trial. Evid Based Complement Alternat Med. 2019 Mar 4;2019:3917282. doi: 10.1155/2019/3917282. eCollection 2019. PMID 30949218